CLINICAL TRIAL: NCT02703246
Title: Tissue Removal During Hysterectomy: The Effect of Vaginal Versus Abdominal Morcellation on Surgical Outcomes
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: investigator left the institution- no plan on having another PI take over
Sponsor: George Washington University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 091553
Record Dates: First submitted 2016-02-08; First posted 2016-03-09 (Estimated); Last update posted 2023-06-05 (Actual); Status verified 2023-06

CONDITIONS: Fibroids
Keywords: Hysterectomy, Vaginal; Hysterectomy, Abdominal
MeSH Terms: conditions — Leiomyoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- abdominal morcellation (Active Comparator): Women randomized to this group will undergo abdominal morcellation.
  Interventions: Procedure: abdominal morcellation
- vaginal morcellation (Active Comparator): Women randomized to this group will undergo vaginal morcellation.
  Interventions: Procedure: vaginal morcellation

INTERVENTIONS:
Procedure: abdominal morcellation — patients will be randomized to receive abdominal morcellation
  Arms: abdominal morcellation
Procedure: vaginal morcellation — patients will be randomized to receive vaginal morcellation
  Arms: vaginal morcellation

SUMMARY:
In this study the investigators will perform a randomized trial to compare the surgical outcomes of vaginal versus abdominal morcellation of the uterus during hysterectomy. In minimally invasive gynecologic surgery small incisions are made in the abdomen and pelvis so that a hysterectomy can be performed by laparoscopy. The challenge is then to remove the uterus, which may be quite large, through these small incisions. One option is to morcellate the uterus and remove the tissue through either a small abdominal incision or an incision in the vagina. When an organ is morcellated it is cut into smaller pieces so that it can be removed, section by section, through a small incision. The investigators will compare these two methods of tissue removal to see whether one results in better surgical outcomes or increased intra-operative or post-operative complications. The primary outcome will be the time it takes to perform the surgery (operative time). Secondary surgical outcomes that will be studied include the amount of blood lost during surgery, post-operative complications, and readmission to the hospital.

DETAILED DESCRIPTION:
Hysterectomy is the most commonly performed non-obstetric procedure in women in the United States, with approximately 400,000 hysterectomies performed each year. Minimally invasive techniques have all been shown to have advantages over laparotomy. These include decreased blood loss, faster recovery time, improved postoperative pain and decreased postoperative complications including wound infections, thromboembolism, iatrogenic injuries and incisional hernias. Due to all of these benefits, the volume of minimally invasive procedures has increased significantly over the last ten years making tissue extraction a widely debated topic.

Morcellation is a technique that allows large pieces of tissue to be removed through small incisions and was originally performed either with a scalpel or manual device until the first power/electric morcellators were introduced in 1993. Since then, power morcellation has made 50,000 to 150,000 minimally invasive hysterectomies possible annually. While the former has been an integral part in the treatment of women with large uteri and uterine fibroids, it has recently come under scrutiny due to multiple concerns including dissemination of undetected malignancy, development of iatrogenic myomas as well as increased number of reported complications and death. This has led the US Food and drug administration in April 2014 to issue a statement discouraging the use of laparoscopic power morcellation.

In the face of the growing bias against electronic mechanical morcellators, other approaches must be investigated and promulgated so that patients may still benefit from minimally invasive gynecologic surgeries. The two commonly used methods for tissue extraction are manual morcellation through mini-laparotomy and vaginal morcellation. In the former, a trocar site enlargement or a new up to 1 inch incision is created through which the specimen is brought to the abdominal surface and morcellated with scalpel.In the latter, tissues are removed in the same fashion but via a colpotomy. The investigators intent is to compare manual morcellation methods (vaginal vs abdominal mini-laparotomy) in order to help surgeons choose the best approach for their patient.

ELIGIBILITY:
Inclusion Criteria:

* Hysterectomy planned for a benign gynecologic reason
* Patient is scheduled to have surgery with one of the minimally invasive gynecologic surgeons at George Washington University Hospital. (Dr. Moawad, Dr. Marfori, or Dr. Vargas)
* Patient is planned for a robotic assisted total laparoscopic hysterectomy (RA-TLH) or a total laparoscopic hysterectomy (TLH)
* Patient is capable of informed consent
* Patient must be between 18 and 65 years of age
* Uterus greater than 12 centimeters in height and 4 centimeters in width or 12 weeks in size

Exclusion Criteria:

* Hysterectomy is indicated for malignancy
* Procedure is anything other than RA-TLH or TLH
* Surgeon is not one of hte minimally invasive surgeons at GWUH
* Surgery is scheduled for a hospital other than GWUH
* Patient does not meet the age requirements.
* Patient is not capable of informed consent
* Uterus is less than 12 cm in heightand 4 cm in width

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-01; Primary Completion 2023-05 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Total operative time | Perioperative
  Time (in minutes) from when first cut is made until last suture is made.

SECONDARY OUTCOMES:
Blood Loss | perioperative
  as measured in cubic centimeters (cc)
Intraoperative complications | perioperative
  Intraoperative complications include: Organ injury (bladder, bowel, vaginal laceration), Estimated Blood Loss>1000cc, and conversion to laparotomy
Post-operative complications | as recorded between end of operation and 4 weeks post operation
  Post-operative complications include: Reoperation, Intensive Care Unit (ICU) admission, Deep Vein Thrombosis/Pulmonary Embolism (DVT/PE), transfusion, Readmission, Bowel obstruction/ileus, Incision seroma/cellulitis/hematoma/separation/hernia, and cuff cellulitis/abcess/dehiscence/granulation tissue

CONTACTS AND LOCATIONS:
Overall Officials: Gaby Moawad, MD, Principal Investigator — George Washington University Medical Faculty Associates
Locations (1):
- George Washington University Medical Faculty Associates, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No